CLINICAL TRIAL: NCT00731978
Title: Near-Infrared Spectroscopy for Intraoperative Restriction of Fluids Trial A Prospective Randomized Study of Near-infrared Spectroscopy Directed Fluid Therapy vs Standard Fluid Therapy in Patients Undergoing Open Elective Colorectal Surgery
Brief Title: NIRF Trial: Near-Infrared Spectroscopy for Intraoperative Restriction of Fluids Trial
Acronym: NIRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hutchinson Technology Inc (Industry)
Responsible Party: BethAnn Guthmueller / Clinical Project Manager, Hutchsinson Technology Incorporated
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H0045
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Colorectal Surgery
Keywords: Near-Infrared Spectroscopy; Intraoperative Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard (No Intervention): Standard intraoperative fluid management
- Restricted (Experimental): Restricted intraoperative fluid management
  Interventions: Procedure: Restricted intraoperative fluid management

INTERVENTIONS:
Procedure: Restricted intraoperative fluid management — Intraoperative fluid management guided by Sto2.
  Other Names: InSpectra StO2
  Arms: Restricted

SUMMARY:
The purpose of this study is to evaluate if the InSpectra StO2 Monitor can safely guide the amount of fluid needed during colorectal surgery.

The study hypothesis is that intraoperative fluid limitation can be safely accomplished when guided by StO2 monitoring, and that this fluid restriction regimen will result in a reduction in postoperative morbidity when compared to standard monitoring and fluid therapy.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective open colorectal surgery
* Age greater than or equal to 18 years
* Low to moderate risk colorectal surgery patients

Exclusion Criteria:

* Unacceptable Baseline vital sign measurements
* High risk colorectal surgery patients
* Jehovah's Witness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Major postoperative complications | within the first 30 days of the postoperative period

SECONDARY OUTCOMES:
StO2 changes during intraoperative fluid management, hospital-free days, surgical site infections, time to first bowel movement, total fluid and total intraoperative fluid volumes, daily fluid volumes through 3 days postoperative, daily weights | within the first 30 days of the postoperative period

CONTACTS AND LOCATIONS:
Overall Officials: Stephen M Cohn, MD, FACS, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - Stanford University School of Medicine, Stanford, California
  - University of Texas Health Science Center (UTHSCSA), San Antonio, Texas